CLINICAL TRIAL: NCT03510325
Title: Sequential Multiple-Assignment Randomized Trials to Compare Antipsychotic Treatments
Brief Title: Sequential Multiple-Assignment Randomized Trials to Compare Antipsychotic Treatments(SMART-CAT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CRC2017ZD03
Record Dates: First submitted 2018-02-12; First posted 2018-04-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia;; Antipsychotics；; first-episode;; switch
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: The sequential multiple assignment randomized trial design (SMART) design is based on the combination of sequential therapy and dynamic therapy, which is more suitable to assess the effectiveness of treatment options in the real world setting. Participants who had an acceptable response to the randomly assigned drug therapy will remain on that treatment for a 12-month treatment period, while non-responders will move to the next phase of the study to receive a new treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- 【Phase 1】 Olanzapine RCT (Experimental): Phase 1 of the trial is a 8-week randomized controlled trial (RCT); patients will be randomly assigned to one of five treatment arms with different oral antipsychotics, one of which is 'Olanzapine RCT'. Non-responders or patients with intolerable side effects in phase 1 will switch to phase 2.
  Interventions: Drug: Phase 1: Olanzapine
- 【Phase 1】 Risperidone RCT (Experimental): Phase 1 of the trial is a 8-week randomized controlled trial (RCT); patients will be randomly assigned to one of five treatment arms with different oral antipsychotics, one of which is 'Risperidone RCT'. Non-responders or patients with intolerable side effects in phase 1 will switch to phase 2.
  Interventions: Drug: Phase 1: Risperidone
- 【Phase 1】 Amisulpride RCT (Experimental): Phase 1 of the trial is a 8-week randomized controlled trial (RCT); patients will be randomly assigned to one of five treatment arms with different oral antipsychotics, one of which is 'Amisulpride RCT'. Non-responders or patients with intolerable side effects in phase 1 will switch to phase 2.
  Interventions: Drug: Phase 1: Amisulpride
- 【Phase 1】 Aripiprazole RCT (Experimental): Phase 1 of the trial is a 8-week randomized controlled trial (RCT); patients will be randomly assigned to one of five 8-week treatment arms with different oral antipsychotics, one of which is 'Aripiprazole RCT'. Non-responders or patients with intolerable side effects in phase 1 will switch to phase 2.
  Interventions: Drug: Phase 1: Aripiprazole
- 【Phase 1】 Perphenazine RCT (Experimental): Phase 1 of the trial is a 8-week randomized controlled trial (RCT); patients will be randomly assigned to one of five treatment arms with different oral antipsychotics, one of which is 'Perphenazine RCT'. Non-responders or patients with intolerable side effects in phase 1 will switch to phase 2.
  Interventions: Drug: Phase 1: Perphenazine
- 【Phase 2】 Olanzapine ESR (Experimental): Non-responders or patients with intolerable side effects in phase 1 will switch to phase 2, a 8-week equipoise-stratified randomization (ESR) trial; patients treated with risperidone, amisulpride, aripiprazole or perphenazine in phase 1 will be randomly assigned to one of three treatment arms, one of which is 'Olanzapine ESR'. Non-responders or patients with intolerable side effects in phase 2 will switch to phase 3.
  Interventions: Drug: Phase 2: Olanzapine
- 【Phase 2】 Amisulpride ESR (Experimental): Non-responders or patients with intolerable side effects in phase 1 will switch to phase 2, a 8-week equipoise-stratified randomization (ESR) trial; patients treated with olanzapine, risperidone, aripiprazole or perphenazine in phase 1 will be randomly assigned to one of three treatment arms, one of which is 'Amisulpride ESR'. Non-responders or patients with intolerable side effects in phase 2 will switch to phase 3.
  Interventions: Drug: Phase 2: Amisulpride
- 【Phase 2】 Clozapine ESR (Experimental): Non-responders or patients with intolerable side effects in phase 1 will switch to phase 2, a 8-week equipoise-stratified randomization (ESR) trial; patients in phase 1 will be randomly assigned to one of three treatment arms, one of which is 'Clozapine ESR'. Non-responders or patients with intolerable side effects in phase 2 will switch to phase 3.
  Interventions: Drug: Phase 2: Clozapine
- 【Phase 3】 Clozapine extended treatment or MECT add-on therapy (Experimental): If a patient received clozapine in phase 2 failed to response, the individual will be assigned to the clozapine extended treatment or modified electroconvulsive therapy (MECT) add-on therapy.
  Interventions: Other: Phase 3A: Clozapine extended treatment or Combined clozapine-MECT therapy
- 【Phase 3】 Clozapine or another SGAs (olanzapine, amisulpride, risperidone, or aripiprazole) (Experimental): Non-clozapine users in phase 2 will be assigned to clozapine or another Second generation antipsychotics (SGAs) not previously used in phase 1 and 2.
  Interventions: Drug: Phase 3B: Clozapine or another SGAs

INTERVENTIONS:
Drug: Phase 1: Olanzapine — Initial dosage: 5-10 mg; recommended dosage: 5-20 mg/d; dosage form: po. duration: 8 weeks
  Arms: 【Phase 1】 Olanzapine RCT
Drug: Phase 1: Risperidone — Initial dosage: 1-2 mg; recommended dosage: 2-6 mg/d; dosage form: po. duration: 8 weeks
  Arms: 【Phase 1】 Risperidone RCT
Drug: Phase 1: Amisulpride — Initial dosage: 200-400 mg; recommended dosage: 400-1200 mg/d; dosage form: po. duration: 8 weeks
  Arms: 【Phase 1】 Amisulpride RCT
Drug: Phase 1: Aripiprazole — Initial dosage: 5-10 mg; recommended dosage: 10-30 mg/d; dosage form: po. duration: 8 weeks
  Arms: 【Phase 1】 Aripiprazole RCT
Drug: Phase 1: Perphenazine — Initial dosage: 2-4 mg; recommended dosage: 6-36 mg/d; dosage form: po. duration: 8 weeks
  Arms: 【Phase 1】 Perphenazine RCT
Drug: Phase 2: Olanzapine — Initial dosage: 5-10 mg; recommended dosage: 5-20 mg/d; dosage form: po. duration: 8 weeks
  Arms: 【Phase 2】 Olanzapine ESR
Drug: Phase 2: Amisulpride — Initial dosage: 200-400 mg; recommended dosage: 400-1200 mg/d; dosage form: po. duration: 8 weeks
  Arms: 【Phase 2】 Amisulpride ESR
Drug: Phase 2: Clozapine — Initial dosage: 25-50 mg; recommended dosage: 200-400 mg/d; dosage form: po. duration: 8 weeks
  Arms: 【Phase 2】 Clozapine ESR
Other: Phase 3A: Clozapine extended treatment or Combined clozapine-MECT therapy — Clozapine extended treatment:
  dosage: 200-600 mg/d; dosage form: po.
  Combined clozapine-MECT therapy:
  Dosage of clozapine: 200-600 mg/d; The modified electroconvulsive therapy (MECT) will be administered three times per week for the first 2 weeks, then twice a week for the next 2 weeks. The total treatment duration is about one month.
  Arms: 【Phase 3】 Clozapine extended treatment or MECT add-on therapy
Drug: Phase 3B: Clozapine or another SGAs — Clozapine:
  Initial dosage: 25-50 mg; recommended dosage: 200-600 mg/d; duration: 8 weeks
  Another Second generation antipsychotics (SGAs) (not previously used in phase 1 and 2): Olanzapine, risperidone, amisulpride, or aripiprazole The dosage of each drug is the same as that of phase 1 and phase 2.
  Arms: 【Phase 3】 Clozapine or another SGAs (olanzapine, amisulpride, risperidone, or aripiprazole)

SUMMARY:
This study is a sequential multiple-assignment randomized trial (RCT) of antipsychotic medication treatment in first-episode schizophrenia patients in the real-world settings.Through analysis of treatment efficacy rate and adverse reactions and pharmacoeconomic evaluation, this project intends to provide evidence for the selection of antipsychotics in FES patients as well as the efficacy and safety of using clozapine in the early phase of schizophrenia treatment by comparing with other SGAs.

DETAILED DESCRIPTION:
A total of 720 first-episode schizophrenia (FES) patients will be enrolled and followed up for 12 months in this study. The trial includes three treatment phases (each phase lasting for 8 weeks) and a naturalistic follow-up phase. Phase 1 is a 8-week randomized controlled trial; patients will be randomly assigned to one of the treatments with oral olanzapine, risperidone, amisulpride, aripiprazole or perphenazine. Patients who had an acceptable response to the randomly assigned drug therapy will remain on that treatment for a 12-month treatment period. Subjects who fail to respond in phase 1 will switch to phase 2, an equipoise-stratified randomization trial, in which patients will be randomly assigned to oral olanzapine, amisulpride or clozapine for another 8 weeks. No-responders in phase 2 will further enter an open label trial (phase 3). Patients who receive clozapine in phase 2 will be assigned to an extended clozapine treatment or modified electroconvulsive therapy add-on therapy (Phase 3A). Patients who were not assigned to clozapine in phase 2 will be assigned to treatment with clozapine or another SGAs not previously used in phase 1 and 2 (Phase 3B).

ELIGIBILITY:
Inclusion criteria:

1. Patients must meet the DSM-5 diagnostic criteria for schizophrenia , schizophreniform disorder or schizoaffective disorder, based upon the structured clinical interview by research psychiatrist using Mini International Neuropsychiatric Interview 7.0 (M.I.N.I. 7.0), review of their clinical records, and input from available informants.
2. Inpatients or outpatients.
3. 16-45 years of age.
4. First episode, and the course no more than 3 years.
5. Drug-naïve, or any antipsychotic medication had been used no more than 2 weeks, and the cumulative antipsychotic drug exposure time no more than 6 weeks in lifetime.
6. The severity of psychotic symptoms is moderate or above, and the specific criteria including: have a score ≥4 on at least one item of Positive and Negative Syndrome Scale (PANSS) (delusions, conceptual disorganization, hallucinatory behavior, grandiosity, or suspiciousness/persecution), and PANSS total score >70.
7. Patients must demonstrate adequate decisional capacity to make a choice about participating in this research study and must provide informed consent to participate.

Exclusion criteria:

1. Patients were excluded if more than 3 years had passed since the onset of psychosis;
2. They met any of the contraindications for any of the study drugs;
3. Mental symptoms were caused by organic disease, severe physical illness, psychoactive substance dependence, mental retardation;
4. They were pregnancy or breast-feeding; they were extreme agitation, stupor or negative suicide.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 762 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy rate | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  A 40% reduction or more of the total score in the Positive and Negative Syndrome Scale (PANSS). The PANSS scale consists of 30 items, and each item is rated on a 7-point scale, ranging from 1 (no symptoms) to 7 (extremely severe).
All-cause dropout rate | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  Marked by the treatment discontinuation for any reasons, including poor efficacy, intolerance of adverse reactions, poor compliance and other reasons.

SECONDARY OUTCOMES:
Change from baseline in Clinician-Rated Dimensions of Psychosis Symptom severity (CRDPS) | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  Clinician-Rated Dimensions of Psychosis Symptom severity (CRDPS). The CRDPS scale evaluates eight symptom dimensions of psychosis. Each symptom domain is rated for the past 7 days on a 5-point scale ranging from 0 (absent) to 4 (present and severe).
Cost inventory | baseline,2 months,4 months, 6 months and 12 months
  Direct medical costs (for example, antipsychotics costs, medical examinations costs, health care and service costs and adverse events costs) and indirect costs (such as traffic, nursing, and losing of labor) of the treatments.
Change from baseline in Clinical Global Impression Scale-Severity (CGI-S) | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  Clinical Global Impression Scale-Severity (CGI-S), including assessment of disease severity and overall efficacy. The severity of the disease was scored on an eight-point scale ranging from 0 (not rated) to 7 (extremely severe). The overall efficacy was assessed on an 8-point scale ranging from 0 (not assessed) to 7 (significant deterioration).
Change from baseline in Calgary Depression Scale for Schizophrenia (CDSS) | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  The Calgary Depression Scale for Schizophrenia (CDSS) consists of nine items, each scored from 0 to 3. A total score greater than 6 is considered depression.
Social function | baseline,2 months,4 months and 6 months and 12 months
  Chinese version of UPSA-B, the UCSD (University of California,San Diego) Performance-based Skills Assessment-Brief, consists of two parts: financial skill (A and B) and communication skill. The score of financial skill A range from 0 to 5. The score of financial skill B range from 0 to 6. The score of communication skill range from 0 to 9. The higher scores mean a better outcome.
Life quality: The Heinirich Quality of life Scale (HRQOL) | baseline,2 months,4 months and 6 months and 12 months
  The Heinirich Quality of life Scale (HRQOL) consists of 21 items, each scored from 0 to 6. The higher scores mean a better outcome.
Life quality: Medication Satisfaction Questionnaire (MSN) | baseline,2 months,4 months and 6 months and 12 months
  Medication Satisfaction Questionnaire (MSN) has one item, scored from 1 to 7. The higher scores indicate higher satisfaction with the medication.
Life quality: Subjective Well-being under Neuroleptics (SWN) | baseline,2 months,4 months and 6 months and 12 months
  Subjective Well-being under Neuroleptics (SWN) consists of 20 items, each scored from 1-6.
Extrapyramidal adverse effects: The Barnes Akathisia Scale (BAS) | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  The Barnes Akathisia Scale (BAS) will be used to evaluate objective performance and subjective experience of akathisia, scored from 0 to 3, and the overall clinical evaluation of akathisia is scored from 0 to 5. The higher scores mean a more serious side effect.
Extrapyramidal adverse effects: Simpson-Angus Extrapyramidal Side Effects Scale (SAS) | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  Simpson-Angus Extrapyramidal Side Effects Scale (SAS) consists of 10 items, each scored from 0 to 4. The higher scores mean a more serious side effect.
Extrapyramidal adverse effects: Abnormal Involuntary Movement Scale (AIMS) | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  Abnormal Involuntary Movement Scale (AIMS) consists of 12 items. The first 10 of 12 items is scored from 0 to 4, and the last 2 is scored from 0 to 1. The higher scores mean the more obvious abnormal involuntary movement.
Sexual dysfunction | baseline,0.5 months,1 months, 2 months,4 months , 6 months , 8 months and 12 months
  Arizona Sexual Experiences Scale (ASEX) includes 5 items, each scored from 1-6. A total score greater than or equal to 19 and any item greater than or equal to 5, or any 3 items greater than or equal to 4, can help clinical diagnosis of sexual dysfunction.
Change from baseline in cognitive function: MCCB | baseline,2 months,4 months and 6 months and 12 months
  MATRICS consensus cognitive battery (MCCB) consists of 10 tests that assess cognitive performance in 7 domains, including processing speed, attention/vigilance, working memory, verbal memory, visual learning, reasoning and problem solving, and social cognition.
Change from baseline in cognitive function: NBSC | baseline,2 months,4 months and 6 months and 12 months
  New cognitive battery for patients with schizophrenia in China(NBSC). NBSC includes 4 tests from MCCB and 5 new tests (Trial making A, BACS, HVLT-R learning and recall, CPTIP, dominant hand Grooved Pegboard, Color Trails I and II, PASAT)
Safety index: Blood pressure | baseline,2 months,4 months and 6 months and 12 months
  Blood pressure in mmHg
Safety index: Heart rate | baseline,2 months,4 months and 6 months and 12 months
  Heart rate
Safety index: Respiratory rate | baseline,2 months,4 months and 6 months and 12 months
  respiratory rate
Safety index: Vital signs | baseline,2 months,4 months and 6 months and 12 months
  body temperature in celsius
Safety index: Blood count | baseline,2 months,4 months and 6 months and 12 months
  Blood count
Safety index: Liver function | baseline,2 months,4 months and 6 months and 12 months
  *Concentration of ALT, AST, GGT, ALP, TB, and DB.
Safety index: renal function | baseline,2 months,4 months and 6 months and 12 months
  *Concentration of serum creatinine, blood urea nitrogen, uric acid, serum cystatin C, homocysteine.
Safety index: thyroid function | baseline,2 months,4 months and 6 months and 12 months
  Thyroid function related hormone levels will be tested, including FT3, FT4, T3, TSH, and T4.
Safety index: prolactin | baseline,2 months,4 months and 6 months and 12 months
  Serum prolactin level
Safety index: QTc interval | baseline,2 months,4 months and 6 months and 12 months
  QTc interval
Metabolic side effects: body weight | baseline,2 months,4 months and 6 months and 12 months
  Weight in kilograms
Metabolic side effects: BMI | baseline,2 months,4 months and 6 months and 12 months
  BMI in kg/m^2
Metabolic side effects: waist circumstance | baseline,2 months,4 months and 6 months and 12 months
  Waist circumstance in centimeter
Metabolic side effects: fasting blood-glucose | baseline,2 months,4 months and 6 months and 12 months
  Fasting blood-glucose
Metabolic side effects: insulin index | baseline,2 months,4 months and 6 months and 12 months
  Insulin resistance was assessed using homeostasis model assessment (HOMA-IR).
Metabolic side effects: serum lipid level | baseline,2 months,4 months and 6 months and 12 months
  Concentration of serum triglyceride, LDL-C(low density lipoprotein cholesterol), HDL-C(high density lipoprotein cholesterol) and apolipoprotein.
Metabolic side effects: assessment of feeding behavior | baseline,2 months,4 months and 6 months and 12 months
  Three-Factor Eating Questionnaire (TFEQ-21) consists of 21 items, including 3 dimensions (non-controlled eating, cognitively restricted eating, and emotional eating). Each item is scored from 1 to 4, and the first 16 item requires reverse scoring before calculating dimension scores. The higher scores mean a higher tendency for non-controlled eating, cognitively restricted eating, and emotional eating.
Metabolic side effects: Visual Analogue Scale (VAS) | baseline,2 months,4 months and 6 months and 12 months
  Visual Analogue Scale (VAS) was used to evaluate the desire to eat, hunger sensation and willingness to eat. The scale consists of 3 items, each scored from 0 to 10. The higher scores mean a stronger desire to eat, hunger sensation and willingness to eat.
Metabolic side effects: Physical Activity Evaluation | baseline,2 months,4 months and 6 months and 12 months
  Physical Activity Evaluation
MRI examinaitons | baseline,2 months and 4 months
  Change of grey matter volume and functional connectivity in certain brain region was focused in the MRI examinations, to evaluate the ability of MRI examinaitons (structural MRI, functional MRI and Magnetic Resonance Spectroscopy) to predict response to antipsychotic treatment in first-episode schizophrenia.
Pharmacogenomics | baseline,2 months,4 months
  *Blood sample was collected and genes related to drug efficacy and adverse reaction were tested to evaluate the ability of pharmacogenomics to predict response to antipsychotic treatment in first-episode schizophrenia.
Lipidomics | baseline,2 months,4 months
  *Serum sample was collected for lipidomic analysis to investigate correlation between serum lipids and rapid weight gain in first-episode schizophrenia.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing Brain Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Dalian Seventh People's Hospital, Dalian, Liaoning
  - Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Seventh People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Guo X, Fan X, Feng T, Wang C, Yao Z, Xu X, Chen Z, Wang H, Xie S, He J, Zhuo K, Xiang Q, Cen H, Wang J, Smith RC, Jin H, Keshavan MS, Marder SR, Davis JM, Jiang K, Xu Y, Liu D. Sequential Multiple-Assignment Randomized Trials to Compare Antipsychotic Treatments (SMART-CAT) in first-episode schizophrenia patients: Rationale and trial design. Schizophr Res. 2021 Apr;230:87-94. doi: 10.1016/j.schres.2020.11.010. Epub 2020 Dec 2. PMID 33279374